CLINICAL TRIAL: NCT04997863
Title: Clinical Efficacy and Safety of Sericin Hydrogel Sheet Impregnated With Bird's Nest Extract in Prevention of Hypertrophic Scar Development at Split-thickness Skin Graft Donor Site
Brief Title: Clinical Efficacy and Safety of Sericin Hydrogel Sheet Impregnated With Bird's Nest Extract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Med Chula IRB 572/64
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Wound; Donor Site Complication; Skin Graft Scar; Scar Conditions and Fibrosis of Skin
Keywords: Sericin; Bird's nest; Hydrogel; Hypertrophic scar; Split-thickness skin graft; Donor site
MeSH Terms: conditions — Wounds and Injuries; Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sericin hydrogel sheet impregnated with EBN extract (Experimental): Apply sericin hydrogel sheet impregnated with EBN extract on one-half of the donor site once daily for 8-12 hours per day for 6 months.
  Interventions: Device: Sericin hydrogel sheet impregnated with EBN extract
- Placebo hydrogel sheet (Placebo Comparator): Apply placebo hydrogel sheet on another half of the donor site once daily for 8-12 hours per day for 6 months.
  Interventions: Device: Placebo hydrogel sheet

INTERVENTIONS:
Device: Sericin hydrogel sheet impregnated with EBN extract — Sericin hydrogel sheet impregnated with EBN extract will be used as a primary dressing for preventing scar development at one-half of the STSG donor site. Then, the donor site will be covered with adhesive tape (secondary dressing). The application of primary and secondary dressings will be done once daily after shower in the morning or evening. Both dressings will be recommended to wear over the donor site for 8-12 hours per day. Patients will be advised to remove both dressings before shower to clean the donor site and the surrounding skin, and then replace them with new wound dressing sheets in the next day. The duration of the dressing application will be 6 months.
  Arms: Sericin hydrogel sheet impregnated with EBN extract
Device: Placebo hydrogel sheet — Placebo hydrogel sheet will be used as a primary dressing for preventing scar development at another half of the STSG donor site. Then, the donor site will be covered with adhesive tape (secondary dressing). The application of primary and secondary dressings will be done once daily after shower in the morning or evening. Both dressings will be recommended to wear over the donor site for 8-12 hours per day. Patients will be advised to remove both dressings before shower to clean the donor site and the surrounding skin, and then replace them with new wound dressing sheets in the next day. The duration of the dressing application will be 6 months.
  Arms: Placebo hydrogel sheet

SUMMARY:
Split-thickness skin graft (STSG) is one of the most common procedures performed in plastic surgery and dermatology. The donor site of skin grafting is expected to heal without scarring. However, hypertrophic scar formation is prevalent among STSG donor sites during scar maturation and has become a significant problem at present. Hypertrophic scar results in aesthetic, physical, functional, and psychological problems, leading to a dramatic impact on patients' quality of life ultimately. There are many current therapeutic approaches for preventing and treating hypertrophic scars; however, they remain clinically unsatisfactory because many treatments have been associated with high recurrent rates, high cost, and side effects. Currently, there are no gold standards for hypertrophic scar therapy. There are many attempts to develop new treatment options for the prevention and management of scarring that are acceptable to both physicians and patients. It has previously been shown that both edible bird's nest (EBN) extract and sericin have effectiveness in reducing scar development. They might be a suitable alternative option for scar prevention and could be used safely. Therefore, the sericin hydrogel sheet impregnated with EBN extract is developed as it is believed that the synergism of these combined compounds would be a great help to prevent the development of scars. This study aims to evaluate the efficacy and safety of sericin hydrogel sheet impregnated with EBN extract for the prevention of scar formation in patients with STSG donor sites.

DETAILED DESCRIPTION:
Prospective, randomized, single-center, double-blinded, placebo-controlled, matched pairs clinical study will be conducted to investigate the efficacy and safety of sericin hydrogel sheet impregnated with EBN extract for the prevention of scar development at STSG donor site. Patients who underwent the STSG procedure at the Division of Plastic and Reconstructive Surgery, Department of Surgery, King Chulalongkorn Memorial Hospital will be considered for inclusion and exclusion criteria. Thirty patients will be enrolled in this study. After complete epithelialization, each donor site will be equally divided into two halves: upper and lower halves. Both halves of the donor site will be randomized into sericin hydrogel sheet impregnated with EBN extract group (treatment group) or placebo hydrogel sheet group (control group). The application of both dressings will be done once daily by the patient in the morning or evening after shower. Both dressings will be recommended to wear over the donor site for 8-12 hours per day. The duration of treatment will be six months. Wound quality at 1, 2, 4, and 6 months after starting application will be measured in terms of erythema level, melanin level, transepidermal water loss by using Cutometer® and scar quality (Vancouver scar scale as well as Patient and Observer Scar Assessment Scale). Adverse reactions will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* STSG donor sites freshly closed not more than 1 month after completed epithelialization
* STSG donor sites are at least 5 x 10 cm2 in size.
* STSG donor sites are located on the thigh.
* Donor sites have not been used previously for skin graft harvesting.
* Aged 18-65 years
* Patients who can read and write Thai language
* Willingness to participate
* Signed consent form

Exclusion Criteria:

* Patients with critical illness (such as systemic infection), major acute illness, or chronic medical illness associated with delayed wound healing (such as poor-controlled diabetes mellitus, end-stage renal disease (ESRD), cancer, or immunocompromised diseases)
* Patients with mental disorder
* Patients with active dermatologic conditions such as contractive skin disorders (e.g., scleroderma), psoriasis, or atopic dermatitis
* After completed epithelialization, patients who used other topical agents or dressings on STSG donor sites within 14 days prior to enrollment
* Known sensitivity or allergy to sericin, EBN, other constituents in hydrogel sheet, or adhesive tape
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar Scale (VSS) score | 6 months
  Clinicians will evaluate scar quality using VSS at 6 months after commencing the dressing application. The range of score is 0 to 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) score | 6 months
  Clinicians will evaluate scar quality using POSAS at 1, 2, 4, and 6 months after commencing the dressing application. The range of score is 1 to 10. Normal skin will be recorded as scale 1. Higher scores mean a worse outcome.
Melanin level | 6 months
  Melanin level will be measured using Cutometer® with mexameter mode at 1, 2, 4, and 6 months after commencing the dressing application.
Erythema level | 6 months
  Erythema level will be measured using Cutometer® with mexameter mode at 1, 2, 4, and 6 months after commencing the dressing application.
Transepidermal water loss (TEWL) | 6 months
  TEWL will be measured using Cutometer® with tewameter mode at 1, 2, 4, and 6 months after commencing the dressing application.
Adverse events | 6 months
  Adverse events resulted from dressing application will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Ph.D, Principal Investigator — Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand